CLINICAL TRIAL: NCT07280949
Title: Comparison of Posterior Transversus Abdominis Plane Block Combined With Sacral Multifidus Plane Block Versus Posterior Transversus Abdominis Plane Block for Laparoscopic Colorectal Surgery: A Randomized Controlled Trial
Brief Title: Posterior Transversus Abdominis Plane Block Combined With Sacral Multifidus Plane Block Versus Posterior Transversus Abdominis Plane Block for Laparoscopic Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nagy Malak , MD, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-318-2025
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Posterior Transversus Abdominis Plane Block; Sacral Multifidus Plane Block; Laparoscopic Colorectal Surgery
Keywords: transversus abdominis plane block; Sacral block; Laparoscopic; Colorectal surgeries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMPB & TAP Block Group (ST-Group): bilateral ultrasound-guided SMPB & TAP block (Active Comparator): Patient in lateral position. A curvilinear ultrasound probe (5-7 MHz) will be placed longitudinally in midline just above median sacral crest. After identifying hyper echoic median sacral crest with overlying hypo echoic latissimus dorsi muscle, the probe will be moved laterally to identify intermediate crest, dorsal sacral foramina (DSF), longissimus thoracic muscle, and multifidus muscle (MFM).
  After optimizing the image at S2 level, 21G 80 mm block needle will be advanced in plane approach until needle reached sacral foramen. A distinct loss of resistance will be felt once the needle pierced the fibrous covering of S2 foramen. After negative aspiration, a total of 20 mL bupivacaine 0.1875% ( 0.19%) will be injected in incrementally, aspirating every 5 ml and the block will be repeated on the other side.
  Interventions: Procedure: sacral multifidus plane block; Procedure: TAP Block: posterior approach
- TAP block Group (T-Group): this group will receive bilateral ultrasound-guided TAP block (Experimental): Technique of TAP Block: posterior approach The patient in semi-lateral position. A linear ultrasound probe (4-12MHz) will be placed posterior to the mid-axillary line between the costal margin and the iliac crest. When scanning posteriorly, transversus abdominis tailed off and turned into aponeurosis. Subsequently, a blunt-ended needle will be introduced into the TAP between the internal oblique and transversus abdominis, posterior to the mid-axillary line and near the aponeurosis. After confirmation with saline solution into the facial plane, as the appearance of a hypo echoic ellipsoid with well-defined margins on ultrasound imaging. After negative aspiration, a total of 20 mL bupivacaine0.1875% ( 0.19%) will be injected in incrementally, aspirating every 5 ml and the block will be repeated on the other side.
  Interventions: Procedure: TAP Block: posterior approach

INTERVENTIONS:
Procedure: sacral multifidus plane block — The patient in lateral position. A curvilinear ultrasound probe (5-7 MHz) will be placed longitudinally in the midline just above the median sacral crest. After identifying the hyper echoic median sacral crest with the overlying hypo echoic latissimus dorsi muscle, the probe will be moved laterally to identify the intermediate crest, the dorsal sacral foramina (DSF), longissimus thoracic muscle, and multifidus muscle (MFM). After optimizing the image at the S2 level, a 21G 80 mm block needle will be advanced in an in plane approach until the needle reached the sacral foramen. A distinct loss of resistance will be felt once the needle pierced the fibrous covering of S2 foramen. After negative aspiration, a total of 20 mL bupivacaine 0.1875% ( 0.19%) will be injected in incrementally, aspirating every 5 ml and the block will be repeated on the other side
  Arms: SMPB & TAP Block Group (ST-Group): bilateral ultrasound-guided SMPB & TAP block
Procedure: TAP Block: posterior approach — The patient in semi-lateral position. A linear ultrasound probe (4-12MHz) will be placed posterior to the mid-axillary line between the costal margin and the iliac crest. When scanning posteriorly, transversus abdominis tailed off and turned into aponeurosis. Subsequently, a blunt-ended needle will be introduced into the TAP between the internal oblique and transversus abdominis, posterior to the mid-axillary line and near the aponeurosis. After confirmation with saline solution into the facial plane, as the appearance of a hypo echoic ellipsoid with well-defined margins on ultrasound imaging. After negative aspiration, a total of 20 mL bupivacaine0.1875% ( 0.19%) will be injected in incrementally, aspirating every 5 ml and the block will be repeated on the other side.

SUMMARY:
The aim of this study is to compare perioperative analgesic efficacy and safety profile of combined SMPB and posterior TAP block versus posterior TAP block in patients undergoing laparoscopic colorectal cancer surgery.

DETAILED DESCRIPTION:
On arrival of the patients to operating room, patients will be secured with 20 gauge intravenous cannula. Monitoring will include ECG, non-invasive arterial blood pressure (NIBP), and pulse oximeter (SpO2). Before receiving general anesthesia, patients will be randomly assigned into one of the two study groups; SMPB with TAP block Group and TAP block Group.

Induction of general anesthesia will be induced with patients after adequate preoxygenation using 1 µg/kg fentanyl (based on lean body weight), 2 mg/kg of propofol (based on total body weight) and 0.5 mg/kg of atracurium (based on the ideal body weight), in addition to 8mg IV dexamethasone for prevention of postoperative nausea & vomiting. Endotracheal intubation will be established. Anesthesia will be maintained by 1.2% MAC of isoflurane with oxygen (50%) in air and 0.1 mg/kg of atracuri¬um will be administered every 20 minutes as main¬tenance anesthetic drugs. Volume-controlled ventilation will be maintained with a tidal volume of 6 mL/kg of ideal body weight and the respiratory rate will be adapted to maintain ET CO2 between 30 and 40 mmHg. Moni¬toring through ECG, NIBP, pulse oximeter and capnograph (ETCO2) continued throughout the surgeries.

US (Siemens ACUSON X300 Ultrasound System) guided blocks will be administered immediately after the induction of anesthesia and prior to surgical incision by consultant anesthesiologist who had experience in regional anesthesia and were familiar with the SMPB & TAP blocks. To achieve double blinding, patients will receive the block by the anesthetist. Another doctor not involved in the block procedure will evaluate the patients intraoperative and postoperative.

SMPB & TAP Block Group (ST-Group): this group will receive bilateral ultrasound-guided SMPB & TAP block TAP block Group (T-Group): this group will receive bilateral ultrasound-guided TAP block Technique of SMPB block: sacral foramen injection technique The patient in lateral position. A curvilinear ultrasound probe (5-7 MHz) will be placed longitudinally in the midline just above the median sacral crest. After identifying the hyper echoic median sacral crest with the overlying hypo echoic latissimus dorsi muscle, the probe will be moved laterally to identify the intermediate crest, the dorsal sacral foramina (DSF), longissimus thoracic muscle, and multifidus muscle (MFM). After optimizing the image at the S2 level, a 21G 80 mm block needle will be advanced in an in plane approach until the needle reached the sacral foramen. A distinct loss of resistance will be felt once the needle pierced the fibrous covering of S2 foramen. After negative aspiration, a total of 20 mL bupivacaine 0.1875% ( 0.19%) will be injected in incrementally, aspirating every 5 ml and the block will be repeated on the other side(15) Technique of TAP Block: posterior approach The patient in semi-lateral position. A linear ultrasound probe (4-12MHz) will be placed posterior to the mid-axillary line between the costal margin and the iliac crest. When scanning posteriorly, transversus abdominis tailed off and turned into aponeurosis. Subsequently, a blunt-ended needle will be introduced into the TAP between the internal oblique and transversus abdominis, posterior to the mid-axillary line and near the aponeurosis. After confirmation with saline solution into the facial plane, as the appearance of a hypo echoic ellipsoid with well-defined margins on ultrasound imaging. After negative aspiration, a total of 20 mL bupivacaine0.1875% ( 0.19%) will be injected in incrementally, aspirating every 5 ml and the block will be repeated on the other side(16).

The surgery can begin after 15 minutes from block time which is the usual time for sterilization.

Intraoperative inadequate analgesia, indicated by increase of heart rate (HR) or mean arterial blood pressure (MAP) more than 20% above preinduction baseline values, will be managed using incremental 50 microgram doses of fentanyl with a maximum total dose of 5 mcg/kg if additional doses are required. Intraoperative fentanyl consumption will be calculated. All patients will receive 10 minutes before the end of surgery 1 mg granisetron or 4 mg ondansetron IV for antiemetic prophylaxis and ketorolac 30mg IV and paracetamol 1g for postoperative analgesia. At the end of surgery, muscle relaxant will be reversed using neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Awake Extubation will be established after adequate reversal of neuromuscular block.

Patients will be transported to post-anesthesia care unit (PACU). In the PACU, patients will be placed in the semi-sitting position, and oxygen will be given via a nonrebreathing facemask with a reservoir bag. Postoperative pain will be assessed using VAS (where 0 corresponds to no pain and 100 mm to the worst pain) at 2, 4, 6, 12, 18, 24 hours postoperatively and on hospital discharge Postoperatively, in the ward, all patients will receive regular analgesia 1 g paracetamol every 6 h, 30 mg ketorolac every 6 h, 1 mg granisetron or 4 mg ondansetron IV for postoperative nausea and vomiting and diphenhydramine 25-50 mg IV for the treatment of pruritus as needed. Intravenous rescue morphine 2 mg if needed will be carried out at patient wake-up to achieve pain control (VAS ≤ 30mm) by an attending anesthesiologist blinded to group allocation. Patients with a VAS score of ≥ 40mm and patients who will request rescue analgesia will be treated with IV morphine in 2 mg increments every 5 minutes with no upper limit for the total administered dose and total morphine consumption will be recorded. If the patient appeared sedated (Ramsay sedation scale > 2), and/or severe morphine-related side effects are encountered including respiratory depression (Spo2 < 95% and/or respiratory rate < 12 breaths/min), allergic reaction, hypotension, or severe pruritus, morphine titration will be stopped and the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Male or female
* ASA class I to III
* Elective laparoscopic or robotic colorectal surgery with or without resections requiring perineal incisions.

Exclusion Criteria:

* Patient refusal
* History of previous abdominal surgery, preoperative bowel obstruction symptoms, and requirement for emergency surgery
* Conversion to open laparotomy
* Coagulopathy, infection at the injection site, allergy to local anesthetics, body mass index > 30 kg/m2, severe hepatic or renal disease, severe cardiopulmonary disease (≥ ASA IV), diabetic or other neuropathies, patients receiving opioids for chronic analgesic therapy, inability to comprehend visual analogue scale (VAS) and patients transferred to the intensive care unit (ICU) post-surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain score (VAS) | 2 hours
  (VAS) at rest and during coughing at 2hr postoperative.

SECONDARY OUTCOMES:
Fentanyl consumption | 6 hours
  Intraoperative fentanyl consumption
Time to first postoperative analgesic request | 24 hours
  Time to first postoperative analgesic request
Total morphine requirements | 24 hours
  Total morphine requirements 24 hours postoperatively
Visual analogue pain score (VAS) | 24 hours
  10. Visual analogue pain score (VAS) at rest and during coughing at 4, 6, 12, 18 and 24 hours postoperatively
Quality of Recovery (QoR-15) scale | 24 hours
  Quality of Recovery (QoR-15) scale at 24 hours after surgery.
Incidence of complications | 24 hours
  Incidence of complications related to the blocks.(infection, hematoma ,bleeding, nerve injury, local anesthetic toxicity, intravascular injection)
Incidence of postoperative nausea and vomiting | 24 hours
  Incidence of postoperative nausea and vomiting (Nausea was recorded on a graded scale, with 0 indicating no symptom, 1 indicating symptoms, 2 indicating symptoms requiring treatment, and 3 indicating a vomiting event
Time to first flatus & development of postoperative ileus | 24 hours
  Time to first flatus & development of postoperative ileus

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided